CLINICAL TRIAL: NCT06393322
Title: Randomized Trial to Evaluate the Usefulness of Mental Health e-Learning
Brief Title: Evaluate the Usefulness of Mental Health e-Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Levinson_AFP
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Depression; Anxiety
Keywords: Depression; Mental Health; Mental Health Literacy; e-Learning; Knowledge; Stigma; Randomized Controlled Trial
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Depression e-Learning A (Experimental)
  Interventions: Other: Depression e-Learning A
- Anxiety e-Learning A (Experimental)
  Interventions: Other: Anxiety e-Learning A
- Depression e-Learning B (Experimental)
  Interventions: Other: Depression e-Learning B
- Anxiety e-Learning B (Experimental)
  Interventions: Other: Anxiety e-Learning B

INTERVENTIONS:
Other: Depression e-Learning A — Participants in Depression e-Learning A will be provided e-learning about depression, consisting of following components:
  1. One multimedia e-learning lesson on depression;
  2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  1. One multimedia e-learning lesson on depression; 2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  Arms: Depression e-Learning A
Other: Depression e-Learning B — Participants in Depression e-Learning B will be provided e-learning about depression, consisting of following components:
  1. One multimedia e-learning lesson on depression;
  2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  1. One multimedia e-learning lesson on depression; 2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  Arms: Depression e-Learning B
Other: Anxiety e-Learning A — Participants in Anxiety e-Learning A will be provided e-learning about anxiety, consisting of following components:
  1. One multimedia e-learning lesson on anxiety;
  2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  Arms: Anxiety e-Learning A
Other: Anxiety e-Learning B — Participants in Anxiety e-Learning B will be provided e-learning about anxiety, consisting of following components:
  1. One multimedia e-learning lesson on anxiety;
  2. A series of 4 'micro-learning' emails (2 emails/week) with small segments of content to reinforce the material from the lesson.
  Arms: Anxiety e-Learning B

SUMMARY:
In this proposal, the investigators plan to study the impact of In this proposal, we plan to study the impact of e-learning on mental health literacy and stigma related to anxiety and depression. Participants will be randomized to one of four groups - Depression e-Learning A, Depression e-Learning B, Anxiety e-Learning A, and Anxiety e-Learning B. All participants will be given access to all e-learning at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Live in Canada
* 45 years of age and over
* Good command of the English language
* Access to email and high speed internet
* Comfortable using email and internet

Exclusion Criteria:

* Lives outside of Canada
* Not 45 years of age or over
* Does not speak English,
* Does not have access to email or high speed internet
* Is not comfortable using email of internet

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Depression Literacy Questionnaire | 0, 2, 4 weeks
  The Depression Literacy Questionnaire assesses mental health literacy specific to depression. The questionnaire consists of 22 items which are true or false. Respondents can answer each item with one of three options - true, false, or I don't know. Each correct response receives one point. Higher scores indicate higher depression literacy.
Change from baseline in the Anxiety Literacy Questionnaire | 0, 2, 4 weeks
  The Anxiety Literacy Questionnaire assesses mental health literacy specific to anxiety. The questionnaire consists of 22 items which are true or false. Respondents can answer each item with one of three options - true, false, or I don't know. Each correct response receives one point. Higher scores indicate higher depression literacy.

SECONDARY OUTCOMES:
Change from baseline in the Depression Stigma Scale | 0, 2, 4 weeks
  The Depression Stigma Scale is a 9-item assessment designed to measure stigma associated with depression with two subscales: personal and perceived. The Personal Stigma Subscale measures stigma in the respondents' own attitudes towards depression by asking them to indicate how strongly they personally agree with nine statements about depression. The Perceived Stigma Subscale measures the respondent's perception about the attitudes of others towards depression by asking them to indicate what they think most other people believe about the same nine statements. Responses to each item are measured on a five-point scale (ranging from zero 'strongly disagree' to four 'strongly agree'). Higher scores indicate higher levels of depression stigma.
Change from baseline in the Generalized Anxiety Stigma Scale | 0, 2, 4 weeks
  The Generalised Anxiety Stigma Scale is analogous, but designed to measure stigma associated with anxiety disorders. It has two subscales: personal and perceived. The Personal Stigma Subscale measures stigma in the respondents' own attitudes towards anxiety disorders by asking them to indicate how strongly they personally agree with 10 statements about anxiety disorders. The Perceived Stigma Subscale measures the respondent's perception about the attitudes of others towards anxiety disorders by asking them to indicate what they think most other people believe about the same 10 statements. Responses to each item are measured on a five-point scale (ranging from zero 'strongly disagree' to four 'strongly agree'). Higher scores indicate higher levels of anxiety stigma.
Participant satisfaction | 2 weeks
  A custom satisfaction questionnaire data adapted from the Information Assessment Method For All (IAM4all) will be collected and saved to assess satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No